CLINICAL TRIAL: NCT01874197
Title: Branched Thoracic Endovascular Grafts for the Treatment of Thoraco-abdominal Aortic Aneurysms: an Investigator-Initiated Study
Brief Title: Branched Thoracic Endovascular Grafts for the Treatment of Thoraco-abdominal Aortic
Acronym: B-TEVAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Matthew P. Sweet, Associate Professor, Surgery, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004379
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2023-05

CONDITIONS: Thoracoabdominal Aortic Aneurysm, Without Rupture
Keywords: Thoracoabdominal Aortic Aneurysm; Branched vessels
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- B -TEVAR (Other): Implantation of the B-TEVAR device
  Interventions: Device: B-TEVAR device

INTERVENTIONS:
Device: B-TEVAR device — Implantation of the Branched Thorcoabdominal aortic anerysm device

SUMMARY:
An investigator-initiated, prospective, consecutively enrolling, non-randomized single institution clinical evaluation of the safety and effectiveness of branched and fenestrated-branched endovascular stent grafts to preserve branch vessels when used in the treatment of patients with thoraco-abdominal aortic aneurysms. The study evaluates non-FDA-approved off the shelf and custom made branched and fenestrated-branched stent grafts manufactured by Cook Medical.

The primary objectives of this study are to determine whether fenestrated-branched and branched endovascular grafts are a safe and effective method of treating patients with thoraco-abdominal aortic aneurysms.

DETAILED DESCRIPTION:
A branched thoracic endograft is a commercially manufactured endograft that has reinforced fenestrations or branches in the graft through which covered stent grafts can be deployed to preserve blood flow into visceral branch vessels.

The branched stent graft is deployed to reline the peri-visceral abdominal aorta. Proximal and distal fixation and seal can be achieved using the branched device, additional Cook Alpha Thoracic devices and/or the Cook Zenith® Flex® device depending on the aortic anatomy.

Once the aortic stent grafts are deployed, the branches are then created. Wires and catheters are used to cross through the reinforced fenestrations into the target visceral arteries. Covered stents are then deployed to extend from the modified aortic graft to the target vessel. The branch stents must create a hemostatic seal with the main endograft as these branches will be constructed within the aneurysm sac. Single or multiple stents may be required for any given branch.

ELIGIBILITY:
Inclusion Criteria:

All patients must meet all of the following inclusion criteria to be eligible for enrollment into this study:

1. Patient is > 18 years of age
2. Patients who are male or non-pregnant female (females of child bearing potential must have a negative pregnancy test prior to enrollment into the study)
3. Patient or Legally Authorized Representative has signed an Institutional Review Board (IRB) approved Informed Consent Form
4. Patient is considered by the treating physician to be at high risk of open surgical repair due to one or more major medical co-morbidities (i.e. CAD, CHF, COPD, CRI, advanced age, generalized deconditioning, or other.) with ASA of 3 or more.
5. The patient has a life expectancy of greater than 1 year.
6. The patient has a thoraco-abdominal aortic aneurysm where necessary visceral branch vessels (i.e. the celiac, superior mesenteric, inferior mesenteric, renal and/or dominant spinal arteries) arise from the aneurysm or seal zones necessary for on-label thoracic endovascular repair
7. Patient has a thoraco-abdominal aortic aneurysm that meets at least one of the following:

   * aneurysm > 5.5 cm in diameter
   * aneurysm has increased in size by 0.5 cm in last 6 months
   * aneurysm is believed to be causing symptoms
8. Patient has sufficient arterial access (femoral and/or iliac) that will allow delivery of the endovascular device with or without the use of a surgical conduit.
9. Patient has suitable proximal (aorta) and distal (aorta or iliac) arteries to allow for adequate fixation and seal:

A. Non-aneurysmal proximal aortic seal zone:

1. with a length of 25 mm of proximal seal in non-aneurysmal aorta, with or without coverage of the left subclavian artery,
2. with an outer wall diameter of no less than 20 mm and no greater 38mm, and

   B. Non-aneurysmal distal aortic or iliac landing zone:
3. With a length of at least 15 mm,
4. Aortic seal zone no less than 15 mm and no greater than 38 mm or Iliac seal zone with an outer wall diameter of no less than 8 mm and no greater than 23 mm.

10. The patient has no more than 5 necessary visceral arteries that require flow preservation.

11. All target visceral artery seal zones are > 4 mm in diameter. 12. Patient must be willing to comply with all required follow-up exams.

Exclusion Criteria:

Patients that meet ANY of the following are not eligible for enrollment into the study:

1. Patient has an active systemic infection
2. Patient has a mycotic aneurysm.
3. Patient has a known hypersensitivity to contrast media that is not amenable to pre-treatment.
4. Patient has an absolute contra-indication to anticoagulation
5. Patient has a known allergy or intolerance to stainless steel, nickel, or gold
6. Patient has a body habitus that would inhibit adequate X-ray visualization of the aorta
7. Patient has a dominant artery to the spinal cord arising from an area of stent graft coverage that is not amenable to preservation using an endovascular branch
8. Patient is currently participating in another investigational device or drug clinical trial
9. Patient has other medical, social or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.
10. Patient has a freely ruptured TAAA with hemodynamic instability
11. Patient has unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina)
12. Patient has had a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned within 30 days of the TAAA repair. Adjunctive procedures for treatment of the TAAA (i.e. carotid-subclavian bypass or iliac conduit) are acceptable.
13. Patient has a history of connective tissue disease (e.g. Marfan or Ehlers Danlos syndromes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2012-08; Primary Completion 2025-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of multi-branched endovascular grafts will be determined by evaluating the proportion of patients that achieve Treatment Success | 12 months post-procedure.

SECONDARY OUTCOMES:
Mortality rates | 12 months

OTHER OUTCOMES:
Technical Success | 12 months
  Technical Success is defined as successful delivery and deployment of the physician modified graft with preservation of unimpeded flow to those branch vessels intended to be preserved.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Sweet, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington/Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data are shared with the Aortic Research Consortium research group

REFERENCES:
- [Background] Aucoin VJ, Motyl CM, Novak Z, Eagleton MJ, Farber MA, Gasper W, Oderich GS, Mendes B, Schanzer A, Tenorio E, Timaran CH, Schneider DB, Sweet MP, Zettervall SL, Beck AW; U.S. Aortic Research Consortium. Predictors and outcomes of spinal cord injury following complex branched/fenestrated endovascular aortic repair in the US Aortic Research Consortium. J Vasc Surg. 2023 Jun;77(6):1578-1587. doi: 10.1016/j.jvs.2023.01.205. Epub 2023 Apr 13. PMID 37059239
- [Background] Chamseddin K, Timaran CH, Oderich GS, Tenorio ER, Farber MA, Parodi FE, Schneider DB, Schanzer A, Beck AW, Sweet MP, Zettervall SL, Mendes B, Eagleton MJ, Gasper WJ; U.S. Aortic Research Consortium. Comparison of upper extremity and transfemoral access for fenestrated-branched endovascular aortic repair. J Vasc Surg. 2023 Mar;77(3):704-711. doi: 10.1016/j.jvs.2022.10.009. Epub 2022 Oct 17. PMID 36257344
- [Background] Zettervall SL, Tenorio ER, Schanzer A, Oderich GS, Timaran CH, Schneider DB, Eagleton M, Farber MA, Gasper WJ, Beck AW, Sweet MP; U.S. Fenestrated and Branched Aortic Research Consortium. Secondary interventions after fenestrated/branched aneurysm repairs are common and nondetrimental to long-term survival. J Vasc Surg. 2022 May;75(5):1530-1538.e4. doi: 10.1016/j.jvs.2021.11.074. Epub 2021 Dec 23. PMID 34954272
- [Background] Tenorio ER, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Parodi FE, Gasper WJ, Beck AW, Sweet MP, Zettervall SL, Huang Y, Oderich GS; U.S. Fenestrated and Branched Aortic Research Consortium. Effect of bridging stent graft selection for directional branches on target artery outcomes of fenestrated-branched endovascular aortic repair in the United States Aortic Research Consortium. J Vasc Surg. 2023 Jul;78(1):10-28.e3. doi: 10.1016/j.jvs.2023.03.025. Epub 2023 Mar 21. PMID 36948277
- [Background] Pujari A, Ahmad M, Sweet MP, Zettervall SL. Overhead arm support reduces radiation exposure during complex endovascular aortic repair. J Vasc Surg. 2023 Apr;77(4):991-996. doi: 10.1016/j.jvs.2022.12.021. Epub 2022 Dec 21. PMID 36565780
- [Background] Edman NI, Schanzer A, Crawford A, Oderich GS, Farber MA, Schneider DB, Timaran CH, Beck AW, Eagleton M, Sweet MP; U.S. Fenestrated and Branched Aortic Research Consortium. Sex-related outcomes after fenestrated-branched endovascular aneurysm repair for thoracoabdominal aortic aneurysms in the U.S. Fenestrated and Branched Aortic Research Consortium. J Vasc Surg. 2021 Sep;74(3):861-870. doi: 10.1016/j.jvs.2021.02.046. Epub 2021 Mar 26. PMID 33775747
- [Background] Sweet MP, Starnes BW, Tatum B. Endovascular treatment of thoracoabdominal aortic aneurysm using physician-modified endografts. J Vasc Surg. 2015 Nov;62(5):1160-7. doi: 10.1016/j.jvs.2015.05.036. Epub 2015 Jul 17. PMID 26194816
- [Background] Timaran CH, Oderich GS, Tenorio ER, Farber MA, Schneider DB, Schanzer A, Beck AW, Sweet MP; Aortic Research Consortium. Expanded Use of Preloaded Branched and Fenestrated Endografts for Endovascular Repair of Complex Aortic Aneurysms. Eur J Vasc Endovasc Surg. 2021 Feb;61(2):219-226. doi: 10.1016/j.ejvs.2020.11.001. Epub 2020 Nov 28. PMID 33262091
- [Background] Schanzer A, Beck AW, Eagleton M, Farber MA, Oderich G, Schneider D, Sweet MP, Crawford A, Timaran C; U.S. Multicenter Fenestrated/Branched Aortic Research Consortium. Results of fenestrated and branched endovascular aortic aneurysm repair after failed infrarenal endovascular aortic aneurysm repair. J Vasc Surg. 2020 Sep;72(3):849-858. doi: 10.1016/j.jvs.2019.11.026. Epub 2020 Mar 3. PMID 32144014
- [Derived] Mesnard T, Huang Y, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Parodi FE, Gasper WJ, Beck AW, Sweet MP, Zetterval SL, Lee A, Oderich GS; United States Aortic Research Consortium. Multicenter Prospective Evaluation of Patient Radiation Exposure During Fenestrated-Branched Endovascular Aortic Repair: A Ten-year Experience. Ann Surg. 2025 Feb 18. doi: 10.1097/SLA.0000000000006676. Online ahead of print. PMID 39963789
- [Derived] Oderich GS, Huang Y, Harmsen WS, Tenorio ER, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Gasper WJ, Beck AW, Sweet MP, Lee WA; United States Aortic Research Consortium. Early and Late Aortic-Related Mortality and Rupture After Fenestrated-Branched Endovascular Aortic Repair of Thoracoabdominal Aortic Aneurysms: A Prospective Multicenter Cohort Study. Circulation. 2024 Oct 22;150(17):1343-1353. doi: 10.1161/CIRCULATIONAHA.123.068234. Epub 2024 Jul 11. PMID 38989575
- [Derived] Finnesgard EJ, Beck AW, Eagleton MJ, Farber MA, Gasper WJ, Lee WA, Oderich GS, Schneider DB, Sweet MP, Timaran CH, Simons JP, Schanzer A; United States Aortic Research Consortium. Severity of acute kidney injury is associated with decreased survival after fenestrated and branched endovascular aortic aneurysm repair. J Vasc Surg. 2023 Oct;78(4):892-901. doi: 10.1016/j.jvs.2023.05.034. Epub 2023 Jun 16. PMID 37330702